CLINICAL TRIAL: NCT06862050
Title: BREATHE Free: Character Strength and Resilience-Based Curriculum for Successful Tobacco Treatment: a Pilot Feasibility Trial
Brief Title: BREATHE Free: a Pilot Feasibility Trial
Acronym: BF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Ban Majeed, Associate Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2051137
Record Dates: First submitted 2025-03-03; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Smoking Cessation; Tobacco Dependence; E-Cig Use; Nicotine Dependence, Other Tobacco Product
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BREATHE Free (Experimental): Attend 12 in-person weekly meetings and go through Breathe Free curriculum.
  Interventions: Behavioral: BREATHE Free Curriculum
- Control (No Intervention): This group will serve as a control group and will receive usual care, referral to tobacco quit line.

INTERVENTIONS:
Behavioral: BREATHE Free Curriculum — Curriculum will teach practices: love, perspective, prudence, hope, humility, forgiveness, spirituality, self-control, teamworking, perseverance, gratitude, and joy.
  Arms: BREATHE Free

SUMMARY:
The overall purpose of this pilot study is to assess the feasibility and acceptability of an in-person faith-based intervention to help people stop tobacco use. The study will address use of different types of tobacco products, such as smoking combustible cigarettes, cigarillos and little filtered cigars, and using/vaping electronic nicotine delivery systems (vape pens, e-cigs, and JUUL).

The intervention consists of 12 weekly meetings in which participants will go through BREATHE Free, a study guide curriculum designed to teach character strengths and promote resilience. This pilot research will provide information and practical lessons on how to improve Breathe Free implementation, increase engagement of the local people, and maximize their benefit.

The main questions it aims to answer are:

* Do participants find BREATHE Free curriculum acceptable, engaging and helpful to stop tobacco use?
* Do participants who complete BREATHE Free curriculum smoke fewer cigarettes per day?

Researchers will assign participants to either BREATHE Free curriculum or usual care.

Participants will:

* Be taught BREATHE Free curriculum or be given information and referral to tobacco quit line
* BREATHE Free group will attend 12 group meetings held on the university campus
* All participants will answer interview questions related to tobacco use, character strengths and resilience
* Expired Carbon Monoxide (CO) will be assessed in all participants.

ELIGIBILITY:
Inclusion Criteria:

* Daily use of one or more tobacco products
* Valid home address in Augusta or the CSRA
* Functioning telephone number
* Speak, read, write in English

Exclusion Criteria:

* Current use of tobacco cessation medications
* Enrolled in tobacco treatment program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Engagement | Weekly assessments, with first assessment in week 2 and last assessment in week 12.
  Active participation in weekly session as reflected by number of weekly accomplishments
Acceptability | Program evaluation will be administered on last meeting (week 12).
  Program evaluation questionnaire will assess, on a 1-5 (ranging from completely disagree - completely agree) scale, participants' attitude and confidence to quit tobacco us.
Acceptability | Program evaluation will be administered on last meeting (week 12).
  Program evaluation questionnaire will assess, on a 1-10 (rated from 1=not at all helpful to 10=extremely helpful) scale, perceived helpfulness of BREATHE Free curriculum in helping participants stop tobacco use.

SECONDARY OUTCOMES:
Average number of cigarette smoked per day | Measured in baseline and weeks 12 and 16
  Number of cigarettes (or cigars) smoked per day (CPD)
Smoking abstinence | Measured in baseline and weeks 12 and 16
  Biochemically verified point prevalence abstinence (7 days)
Resilience | Measured in baseline and weeks 12 and 16
  Connor-Davidson Resilience Scale 10 (CD-RISC-10) score

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided